CLINICAL TRIAL: NCT00310895
Title: A Phase I, Sequential Cohort, Dose Escalation Trial to Determine the Safety, Tolerability, and MTD of GRN163L in Patients With Refractory or Relapsed Solid Tumor Malignancies
Brief Title: Safety and Dose Study of GRN163L Administered to Patients With Refractory or Relapsed Solid Tumor Malignancies
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Geron Corporation (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GRN163L CP05-101
Record Dates: First submitted 2006-04-04; First posted 2006-04-05 (Estimated); Last update posted 2015-12-24 (Estimated); Status verified 2015-12

CONDITIONS: Solid Tumor Malignancies
Keywords: Refractory; Relapsed
MeSH Terms: conditions — Recurrence | interventions — imetelstat

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Dose escalation (Experimental): Treatment Schedule 3 will consist of dosing on Days 1, 4, 8, and 11 of each 21 day cycle (3 weeks equals 1 cycle) and Treatment Schedule 4 will consist of dosing on Day 1 of each 28 day cycle (4 weeks equals 1 cycle)
  Interventions: Drug: Imetelstat Sodium (GRN163L)

INTERVENTIONS:
Drug: Imetelstat Sodium (GRN163L) — Dose increase by 25% if tolerated infused over 2 hours

SUMMARY:
The purpose of this study is to determine the safety and the maximum tolerated dose of GRN163L administration in treating patients with refractory or relapsed solid tumor malignancies.

DETAILED DESCRIPTION:
GRN163L is a telomerase template antagonist with in vitro and in vivo activity in a variety of tumor model systems. Telomerase is an enzyme that is active primarily in tumor cells and is crucial for the indefinite growth of tumor cells. Inhibition of telomerase may result in antineoplastic effects.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Male or female
* Measurable or evaluable solid tumor malignancy
* Relapsed, refractory, locally advanced, or metastatic disease
* Disease refractory to or not amenable to standard therapy
* Karnofsky performance status 70-100%
* Life expectancy 3 months or greater

Exclusion Criteria:

* Pregnant or lactating women
* Primary central nervous system(CNS) malignancy or active CNS metastases
* Hematologic malignancy
* Chemotherapy within 4 weeks prior to study
* Mitomycin C, nitrosoureas within 6 weeks prior to study
* High dose chemotherapy with stem cell support within 6 months prior to study
* Signal transduction inhibitors, monoclonal antibodies, etc. within 4 weeks prior to study
* Systemic hormonal therapy within 4 weeks prior to study
* Anticoagulant therapy, antiplatelet therapy within 2 weeks prior to study
* Radiotherapy within 4 weeks prior to study
* Significant cardiovascular disease
* Serious/active infection
* Major surgical procedures within 2 weeks

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 85 (Estimated)
Dates: Start 2006-03; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Safety, DLT, and MTD | Measured during the first cycle of treatment

SECONDARY OUTCOMES:
PK profile and disease response | Within the first 2 cycles of treatment

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - The University of Chicago Medical Center, Chicago, Illinois
  - Wayne State University, Karmanos Cancer Center, Detroit, Michigan

REFERENCES:
- See also: Related Info — http://www.geron.com